CLINICAL TRIAL: NCT02075723
Title: Effect of Sleep Restriction on Metabolic Disturbances Caused by Overfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, José HABA-RUBIO, MD, University of Lausanne Hospitals
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SleepDep 02/14
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Overfeeding + sleep restriction (Experimental): overfeeding condition (130 % of energy requirements ) + 6 days of sleep restriction (4 hours per night)
  Interventions: Dietary Supplement: Overfeeding (130 % of energy requirements ); Behavioral: Sleep restriction (4 hours per night)
- Overfeeding + normal sleep duration (Experimental): overfeeding condition (130 % of energy requirements ) + 6 days of normal sleep duration (8 hours per night)
  Interventions: Dietary Supplement: Overfeeding (130 % of energy requirements )

INTERVENTIONS:
Dietary Supplement: Overfeeding (130 % of energy requirements ) — Overfeeding (130 % of energy requirements )
Behavioral: Sleep restriction (4 hours per night) — Sleep restriction (4 hours per night)
  Arms: Overfeeding + sleep restriction

SUMMARY:
The purpose of this study is to determine if sleep restriction provokes an increase in risk factors for metabolic diseases, such as elevation of ectopic fat and decreased sensitivity to insulin. We propose to evaluate the effect of sleep restriction in a model of metabolic challenge (overfeeding) caricaturing the conditions of modern societies everyday life .

DETAILED DESCRIPTION:
General hypothesis :

In overfeeding condition, the stress response generated by partial sleep restriction of six days will induce an accumulation of fat in the liver and a decreased insulin sensitivity of adipose tissue , liver and muscle, more pronounced that in overfeeding condition only, provoked by a deregulation of the nocturnal lipolysis .

Specific goals :

Purpose 1 : To measure the accumulation of fat in the liver (measured by nuclear magnetic resonance ) and the tissue insulin sensitivity ( measured by a test meal ) in response to a sleep restriction in overfeeding condition .

Hypothesis 1: In overfeeding condition (130 % of energy requirements ) , hepatic lipid accumulation will be higher after 6 days of sleep restriction (4 hours per night) compared to a control condition (8 hours of sleep per night ) . Decreased sensitivity to insulin in the liver, adipose tissue and the associated muscle will be associated at this ectopic fat accumulation.

Purpose 2 : To determine the alteration of lipolysis in response to sleep restriction in overfeeding condition.

Hypothesis 2: In overfeeding condition, sleep restriction will increase the concentrations of circulating fatty acids and glycerol in relation to condition of normal sleep.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* BMI 18.5-25 kg/m2
* Blood pressure at rest less than 140/ 90 mmHg .
* Physical activity level: sedentary or light (< 3 hours of sport per week )
* Lack of sleep pathology ( including sleep apnea and insomnia )
* Regular sleep-wake cycles
* Average duration of sleep over 7h
* Circadian Typology by Horne & Ostberg questionnaire ≥ 30 and ≤ 70
* Score questionnaire Pittsburgh Sleep Quality Index ≤ 5
* Screening polysomnography showing sleep efficiency ≥ 85 % and apnea- hypopnea index and periodic leg movements < 15 / h .

Exclusion Criteria:

* Current smoking
* Family history of diabetes
* History of sleep disorders
* Circadian Typology by Horne & Ostberg [ 16-30 ] or [ 70-86 ]
* Score questionnaire Pittsburgh Sleep Quality Inde x> 5
* Polysomnography indicating a sleep efficiency <85% and apnea-hypopnea index and periodic leg movements > 15 / h.
* Consumption of more than 3 coffees a day
* Drinking alcool (more than 10g /d)
* Use of Drugs
* Medication
* Night work by shifts
* Average duration of sleep less than 7 hours per night
* Occupational Risks in sleep restriction conditions: e.g. professional drivers
* Special Diet ( vegetarianism, veganism , etc. )
* Change in weight of more than 3 kg in the last 3 months
* Consumption of more than 3 dl sugar-sweetened beverages per day ( sodas, energy drinks , fruit juice , flavored milk sugar )
* Contraindication for magnetic resonance imaging ( pacemaker , previous eye surgery, the presence of metal implant or foreign body, Claustrophobia, etc. )
* For women: pregnancy (current or desired)
* Hemoglobin level < 13.5g/dl for men and < 12.5g/dl for women
* Ferritin level < 50ug / l
* Blood donation in the last 8 weeks

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Accumulation of fat in the liver (measured by nuclear magnetic resonance ) and the tissue insulin sensitivity ( measured by a test meal ) in response to a sleep restriction in overfeeding condition . | After 6 days of sleep restriction (4 h/day) vs. normal sleep (8 h/day)

SECONDARY OUTCOMES:
Blood concentrations of circulating fatty acids and glycerol | After 6 days of sleep restriction (4 h/day) vs. normal sleep (8 h/day)

CONTACTS AND LOCATIONS:
Overall Officials: José Haba-Rubio, MD, Principal Investigator — Center for Investigation and Research on Sleep, University Hospital, Lausanne, Switzerland
Locations (1):
- Center for Investigation and Reseaarch on Sleep and Physiology Department, University Hospital, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Cros J, Pianezzi E, Rosset R, Egli L, Schneiter P, Cornette F, Pouymayou B, Heinzer R, Tappy L, Kreis R, Boesch C, Haba-Rubio J, Lecoultre V. Impact of sleep restriction on metabolic outcomes induced by overfeeding: a randomized controlled trial in healthy individuals. Am J Clin Nutr. 2019 Jan 1;109(1):17-28. doi: 10.1093/ajcn/nqy215. PMID 30615104
- See also: Center for Investigation and Research on Sleep, University Hospital, Lausanne, Switzerland — http://www.chuv.ch/sommeil